CLINICAL TRIAL: NCT00000831
Title: Virologic Responses To New Nucleoside Regimens After Prolonged ZDV or ddI Monotherapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: ACTG 302; 11277 (Registry Identifier: DAIDS ES Registry Number)
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2021-11-04 (Actual); Status verified 2021-10

CONDITIONS: HIV Infections
Keywords: Didanosine; Drug Therapy, Combination; AIDS-Related Complex; Antiviral Agents; Zidovudine; Stavudine; Lamivudine; Drug Combinations
MeSH Terms: conditions — HIV Infections; AIDS-Related Complex | interventions — Lamivudine; Stavudine; Zidovudine; Didanosine

INTERVENTIONS:
Drug: Lamivudine
Drug: Stavudine
Drug: Zidovudine
Drug: Didanosine

SUMMARY:
To elucidate the relationship between virologic risk factors and immunologic and clinical progression in patients receiving monotherapy in protocol ACTG 175, and to compare new treatment regimens with combinations of reverse transcriptase inhibitors in long-term recipients of monotherapy. Specifically, to determine, in patients who have been taking zidovudine (AZT) alone for a long time, whether it is beneficial to add lamivudine (3TC) to AZT or to switch to d4T alone, and also to determine, in patients who have been taking didanosine (ddI) alone for a long time, whether it is beneficial to add AZT or AZT/3TC to ddI.

Characteristics of virus replication, pathogenicity, and resistance are thought to determine the durability of virologic and clinical response to nucleoside reverse transcriptase inhibitors. Previous results of ACTG 175 suggest that either a switch to ddI or addition of ddI in patients receiving AZT results in better clinical, virologic, and CD4 cell response compared to continuation of AZT alone.

DETAILED DESCRIPTION:
Characteristics of virus replication, pathogenicity, and resistance are thought to determine the durability of virologic and clinical response to nucleoside reverse transcriptase inhibitors. Previous results of ACTG 175 suggest that either a switch to ddI or addition of ddI in patients receiving AZT results in better clinical, virologic, and CD4 cell response compared to continuation of AZT alone.

Patients with prior AZT experience only are randomized to receive either d4T alone or AZT/3TC. Patients with prior ddI experience only are randomized to receive ddI/AZT or ddI/AZT/3TC. PER AMENDMENT 8/27/96: The study has been extended 6 months and treatment will be available until March 15, 1997 at the latest. Each patient will have regularly scheduled 12 week safety visits during the extension period.

AS PER AMENDMENT 1/22/97: The study has been extended for approximately 16 additional weeks beyond the current 6-month extension. Subjects will be unblinded to their assigned regimen beginning 2/21/97 and will continue therapy for up to 16 weeks in open-label fashion. AS PER AMENDMENT 5/9/97: The study has been extended for an additional 8 weeks; study drug will not be provided after 9/15/97.

ELIGIBILITY:
Inclusion Criteria

Concurrent Medication:

Recommended:

* PCP prophylaxis in patients with CD4 count <= 200 cells/mm3.

Allowed:

* Chemophylaxis against Mycobacterium tuberculosis.
* Acyclovir.
* Vaccination with pneumococcal vaccine polyvalent.
* Haemophilus B Conjugate vaccine.
* Chemoprophylaxis for MAC and Toxoplasma gondii.
* Antibiotics.
* Recombinant erythropoietin ( EPO ) and G-CSF.
* Systemic corticosteroids for < 21 days.
* Regularly prescribed medications such as antipyretics, analgesics, allergy medications, antidepressants, sleep medications, and oral contraceptives.
* Vitamins and herbal therapies.

Concurrent Treatment:

Allowed:

* Limited local radiation therapy to skin.
* Blood transfusions if 3 units or less per 21-day period.
* Acupuncture.
* Visualization techniques.

Patients must have:

* Completed AZT or ddI monotherapy on ACTG 175 and remained on that regimen during any subsequent interval.
* Not reached an ACTG 175 endpoint prior to May 1, 1995.
* Consent of parent or guardian if less than 18 years old.

PER AMENDMENT 8/27/96:

* Patients must be on study/on treatment at the time the protocol study treatment is extended.

Exclusion Criteria

Co-existing Condition:

Patients with the following symptoms or conditions are excluded:

* Grade 2 or worse peripheral neuropathy.
* Malignancy requiring systemic therapy.

Concurrent Medication:

Excluded:

* Anti-HIV drugs other than study drugs.
* Biologic response modifiers.
* Systemic cytotoxic chemotherapy.
* Any drug known to affect glucuronidation and/or clearance of AZT.

Concurrent Treatment:

Excluded:

* Radiation therapy other than limited local therapy to skin.

Patients with the following prior condition are excluded:

* History of acute or chronic pancreatitis.

Prior Medication:

Excluded:

* Prior 3TC.
* Acute therapy for an infection (other than HIV) or other medical illness within 14 days prior to study entry.

Current ethanol abuse.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 280
Dates: Study Completion 1998-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Katzenstein D, Study Chair; Hammer S, Study Chair
Locations (40):
- United States (38):
  - Alabama Therapeutics CRS, Birmingham, Alabama
  - USC CRS, Los Angeles, California
  - UCLA CARE Center CRS, Los Angeles, California
  - Stanford CRS, Palo Alto, California
  - Ucsd, Avrc Crs, San Diego, California
  - Ucsf Aids Crs, San Francisco, California
  - Santa Clara Valley Med. Ctr., San Jose, California
  - San Mateo County AIDS Program, San Mateo, California
  - Harbor-UCLA Med. Ctr. CRS, Torrance, California
  - University of Colorado Hospital CRS, Aurora, Colorado
  - Univ. of Miami AIDS CRS, Miami, Florida
  - Emory Univ. Hemophilia Program Office, Atlanta, Georgia
  - Northwestern University CRS, Chicago, Illinois
  - Cook County Hosp. CORE Ctr., Chicago, Illinois
  - Rush Univ. Med. Ctr. ACTG CRS, Chicago, Illinois
  - Indiana Univ. School of Medicine, Infectious Disease Research Clinic, Indianapolis, Indiana
  - Tulane Hemophilia Treatment Ctr., New Orleans, Louisiana
  - Johns Hopkins Adult AIDS CRS, Baltimore, Maryland
  - Massachusetts General Hospital ACTG CRS, Boston, Massachusetts
  - Bmc Actg Crs, Boston, Massachusetts
  - Beth Israel Deaconess - East Campus A0102 CRS, Boston, Massachusetts
  - Beth Israel Deaconess Med. Ctr., ACTG CRS, Boston, Massachusetts
  - University of Minnesota, ACTU, Minneapolis, Minnesota
  - St. Louis ConnectCare, Infectious Diseases Clinic, St Louis, Missouri
  - Washington U CRS, St Louis, Missouri
  - Univ. of Nebraska Med. Ctr., Durham Outpatient Ctr., Omaha, Nebraska
  - SUNY - Buffalo, Erie County Medical Ctr., Buffalo, New York
  - NY Univ. HIV/AIDS CRS, New York, New York
  - Cornell University A2201, New York, New York
  - Univ. of Rochester ACTG CRS, Rochester, New York
  - Unc Aids Crs, Chapel Hill, North Carolina
  - Carolinas HealthCare System, Carolinas Med. Ctr., Charlotte, North Carolina
  - Regional Center for Infectious Disease, Wendover Medical Center CRS, Greensboro, North Carolina
  - Univ. of Cincinnati CRS, Cincinnati, Ohio
  - Case CRS, Cleveland, Ohio
  - The Ohio State Univ. AIDS CRS, Columbus, Ohio
  - Hosp. of the Univ. of Pennsylvania CRS, Philadelphia, Pennsylvania
  - University of Washington AIDS CRS, Seattle, Washington
- Puerto Rico-AIDS CRS, San Juan, Puerto Rico
- Mbeya Med. Research Program, Mbeya Referral Hosp. CRS, Mbeya, Tanzania

REFERENCES:
- [Background] Shulman NS, Machekano RA, Shafer RW, Winters MA, Zolopa AR, Liou SH, Hughes M, Katzenstein DA; AIDS Clinical Trials Group 302 Study Team. Genotypic correlates of a virologic response to stavudine after zidovudine monotherapy. J Acquir Immune Defic Syndr. 2001 Aug 1;27(4):377-80. doi: 10.1097/00126334-200108010-00008. PMID 11468426
- [Background] Katzenstein DA, Hughes M, Albrecht M, Hammer S, Para M, Murphy R, Valdez H, Haubrich R, Liou S. Virologic and CD4+ cell responses to new nucleoside regimens: switching to stavudine or adding lamivudine after prolonged zidovudine treatment of human immunodeficiency virus infection. ACTG 302 Study Team. AIDS Clinical Trials Group. AIDS Res Hum Retroviruses. 2000 Jul 20;16(11):1031-7. doi: 10.1089/08892220050075282. PMID 10933617
- [Background] Shulman NS, Hughes MD, Winters MA, Shafer RW, Zolopa AR, Hellmann NS, Bates M, Whitcomb JM, Katzenstein DA. Subtle decreases in stavudine phenotypic susceptibility predict poor virologic response to stavudine monotherapy in zidovudine-experienced patients. J Acquir Immune Defic Syndr. 2002 Oct 1;31(2):121-7. doi: 10.1097/00126334-200210010-00001. PMID 12394789